CLINICAL TRIAL: NCT00861770
Title: Prospective Protocol for Utilizing Blood Volume Measurements in the Treatment of Heart Failure Patients
Brief Title: Utilizing Blood Volume Measurements in the Treatment of Heart Failure Patients
Acronym: TEAM UF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Collaborators: Daxor Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCC28158
Record Dates: First submitted 2009-03-11; First posted 2009-03-13 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Ultrafiltration; Blood Volume Measurement
MeSH Terms: conditions — Heart Failure | interventions — Ultrafiltration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Control (Other): All subjects will receive blood volume measurement immediately before and 30 minutes after ultrafiltration is completed. In the control group, the treating physician will not see the blood volume measurement results and treat according to standard of care.
  Interventions: Other: Ultrafiltration
- 2 - BVM (Experimental): Ultrafiltration will be guided by blood volume measurement results.
  Interventions: Other: Ultrafiltration using BVM

INTERVENTIONS:
Other: Ultrafiltration — Ultrafiltration based on standard of care.
  Arms: 1 - Control
Other: Ultrafiltration using BVM — Ultrafiltration will be guided by blood volume measurement results.
  Arms: 2 - BVM

SUMMARY:
This will be a clinical test to determine if using blood volume measurements (BVM) to help guide fluid removal with ultrafiltration in patients hospitalized with decompensated heart failure leads to improved outcomes.

DETAILED DESCRIPTION:
Subjects will be randomized into two groups. In the control group, the treating physician will not see the blood volume measurement results. In the experimental group, the physician will be given the blood volume measurement results. Ultrafiltration is performed based on the results of blood volume measurement in the experimental group followed by repeat blood volume analysis after 30 minutes of the completion of ultrafiltration. Clinical and laboratory assessment as per the standard of care will be used to assess overall fluid status, and blood volume measurement results will be used as the assessment of intravascular fluid. These assessments will be used to determine a goal quantity of fluid to be removed. All subjects will return for a clinical assessment at 30 and 90 days and laboratory data will be drawn at that time to evaluate renal functional indices, electrolytes and blood volume measurements.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of heart failure
* >/= 2 criteria of volume overload

  1. JVD > 7 cm
  2. Ascites
  3. Lower extremity edema
  4. Sacral Edema
  5. Pleural effusion by clinical or radiologic criteria
* CKD 3 or worse renal function ClCR < 60 ml/min
* HCT < 40%
* Serum Albumin >/= 2.5 gm/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine if using blood volume measurement to help guide fluid removal with ultrafiltration in patients hospitalized with decompensated heart failure leads to improved outcomes. | 90 days
Change in serum creatinine ≥ 0.5 mg/dL. | 30 and 90 days
Symptomatic hypotension during ultrafiltration. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Saltzberg, MD, FACC, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States